CLINICAL TRIAL: NCT00249158
Title: Risperidone in the Treatment of Behavioural and Psychological Signs and Symptoms in Dementia (BPSSD): a Multicentre, Double-blind, Placebo-controlled Parallel-group Trial
Brief Title: A Study of the Effectiveness and Safety of Risperidone in the Treatment of Behavioral Disturbances in Patients With Dementia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag Pty Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006010
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Dementia; Alzheimer Disease; Vascular Dementia
Keywords: Dementia; Alzheimer's Disease; vascular dementia; mixed dementia; risperidone; nursing home
MeSH Terms: conditions — Dementia; Alzheimer Disease; Dementia, Vascular; Mixed Dementias | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
The purpose of the study is to compare the effectiveness of an oral formulation of risperidone (an antipsychotic medication) to that of placebo for treating behavioral and psychological signs and symptoms in dementia (BPSSD), specifically aggression, delusions, and hallucinations, in patients with dementia.

DETAILED DESCRIPTION:
Dementia is a term used for a collection of symptoms that can be caused by a number of diseases or injuries that affect the brain. Individuals with dementia have a loss of function in cognition (thinking, perception, learning, verbal communication, memory, judgment), which may lead to behavioral and personality changes (for example, agitation, delusions, hallucinations). Some causes of dementia are reversible; however, irreversible dementia is caused by certain conditions, such as Alzheimer's disease. Dementia is common in elderly individuals, but it is not a normal part of aging. This is a randomized, double-blind, parallel-group, placebo-controlled study comparing the effectiveness and safety of risperidone to placebo in patients with behavioral disturbances associated with dementia. The study is composed of two periods: a 1-week run-in period in which patients are discontinued from other antipsychotic drugs and take placebo twice daily and a 12-week double-blind period. At the end of the run-in period, patients are randomly assigned to oral solutions of either risperidone or placebo. The starting dose of risperidone is 0.25 mg twice daily and increasing to 0.5 mg twice daily (1 mg/day). If 1 mg/day shows an insufficient response, a maximum of 1 mg twice daily of risperidone is permitted. The patient receives study drugs for the 12-week double-blind period. The primary measure of effectiveness is the change from baseline to the end of double-blind treatment in the Cohen-Mansfield Agitation Inventory (CMAI), a questionnaire evaluating agitation. Additional measures of efficacy include the change from baseline to end of double-blind treatment in the Behavior Pathology in Alzheimer's Disease Rating Scale (BEHAVE-AD), a rating scale used to evaluate behavior symptoms in patients with Alzheimer's disease; the Clinical Global Impressions (CGI), a rating system used to evaluate the overall and severity of clinical change in a patient with various diseases affecting the brain; the Functional Assessment Staging (FAST), a diagnosis tool for determining the stage of dementia; and the Mini-Mental State Examination (MMSE), a clinical measure used to evaluate cognition. Safety evaluations include the incidence of adverse events; results of clinical laboratory tests (hematology and biochemistry); measurements of vital signs and body weight; physical examination findings; and the Extrapyramidal Symptoms Rating Scale (ESRS), a scale used to measure effects of antipsychotic medications on motor functions of the patient. The study hypothesis is that risperidone is more effective than placebo, as measured by the total aggression score on the CMAI, in treating behavioral disturbances in demented patients. Risperidone oral solution (1 mg/mL). Starting doses of 0.25 mg twice daily and increasing to 0.5 mg twice daily (1 mg/day). If 1 mg/day shows an insufficient response, a maximum of 1 mg twice daily of risperidone is permitted. Total treatment duration is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Dementia of the Alzheimer's type with behavioral disturbance, vascular dementia with behavioral disturbance, or mixed dementia, as classified by DSM-IV (the Diagnostic and Statistical Manual of Mental Diseases, 4th edition)
* a score >=4 on the FAST (Functional Assessment Staging, a diagnosis tool for determining the stage of dementia) and a score <=23 on the MMSE (Mini-Mental State Examination, a clinical measure used to evaluate cognition)
* a BEHAVE-AD (Behavior Pathology in Alzheimer's Disease Rating Scale) total score >=8, and a BEHAVE-AD global rating >=1
* patient must be living in an nursing home for >=1 month. Exclusion Criteria:
* Patients with other medical or neurological conditions other than dementia in which cognition is diminished (for example, severe anemia, severe liver, heart, lung, and kidney malfunctions, Parkinson's disease)
* diagnosis of depression within the 6 months before study entry, schizophrenia, bipolar affective disorder, or schizoaffective disorder
* history of or moderate to severe tardive dyskinesia, (a condition of uncontrollable movements of the tongue, lips, face, trunk, hands and feet that is seen in patients receiving long-term medication with certain types of antipsychotic drugs)
* abnormal clinical laboratory test findings.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 1998-03; Study Completion 2001-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the end of double-blind treatment in total aggression score of the CMAI (Cohen-Mansfield Agitation Inventory).

SECONDARY OUTCOMES:
Change from baseline to end of double-blind treatment in global and total BEHAVE-AD score, BEHAVE-AD cluster scores and in CMAI cluster scores, CGI, and in FAST MMSE; safety evaluations conducted throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Pty Ltd Clinical Trial, Study Director — Janssen-Cilag Pty Ltd

REFERENCES:
- [Result] Brodaty H, Ames D, Snowdon J, Woodward M, Kirwan J, Clarnette R, Lee E, Lyons B, Grossman F. A randomized placebo-controlled trial of risperidone for the treatment of aggression, agitation, and psychosis of dementia. J Clin Psychiatry. 2003 Feb;64(2):134-43. doi: 10.4088/jcp.v64n0205. PMID 12633121